CLINICAL TRIAL: NCT04909554
Title: MRI-based Approaches for Multi-parametric Model to Early Predict Pathological Complete Response to Neoadjuvant Chemotherapy in Breast Cancer (NeoMDSS)
Brief Title: MRI-based Approaches for Multi-parametric Model to Early Predict Pathological Complete Response to Neoadjuvant Therapy in Breast Cancer
Acronym: NeoMDSS
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shantou Central Hospital (Other); The First Affiliated Hospital of Clinical Medicine of Guangdong Pharmaceutical University (Unknown); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Other Study IDs: 20210504
Record Dates: First submitted 2021-05-09; First posted 2021-06-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Magnetic resonance imaging (MRI); Neoadjuvant therapy (NAT); therapeutic response; breast cancer; early prediction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the training cohort: From January 2019 to December 2020, 140 patients from Guangdong Province People's Hospital with complete clinicopathological information and available images of MRI before treatment and after 1st-NAT were retrospectively recruited for the training cohort
- the internal validation cohort: From June 2021 and December 2023, 120 patients from Guangdong Province People's Hospital were prospectively recruited for the internal validation cohort.
- the external validation cohort: From June 2021 and December 2023, 41 patients from Shantou Central Hospital, The First Affiliated Hospital of Guangdong Pharmaceutical University and The First People's Hospital of Foshan were prospectively recruited for the external validation cohort.

SUMMARY:
The purpose of this clinical research is to evaluate the accuracy of a multi-parametric model based on magnetic resonance imaging (MRI) in predicting pathological complete response (pCR) after the first cycle of neoadjuvant therapy (NAT) given to patients with locally advanced breast cancer, thus allowing early chemotherapy regimen modification to increase number of patients achieving pCR or save patients from toxic effects of ineffective chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent cancer among women worldwide. NAT has been well established in managing breast cancer for patients with locally advanced cancer and early-stage operable breast cancers of specific molecular subtypes. Though pCR has been demonstrated to be associated with better survival, it can only be judged by pathological testing of surgically resected specimens. Thus, predicting pCR earlier during NAT is imperative and can timely switch to a new personalized treatment strategy and exempt from unnecessary chemotherapy toxicity for patients.

This is a multicenter, prospective cohort study of 301 patients undergoing MRI after the first cycle of neoadjuvant chemotherapy. This project plans to establish and validate a model for determining pCR during NAT in breast cancer based on clinical information, imaging and pathological information of patients in multiple centers, in order to provide important references for further early diagnosis and personalized treatment.

1. Collecting MRI images data, clinical and pathological information, treatment regimens, and curative effect information to build an MRI-based, multi-parametric model.
2. Evaluating the performance of model through internal and external validation cohort by using the receiver operating characteristic (ROC) curve, the area under the curve (AUC), discrimination and calibration measures.

ELIGIBILITY:
1. For training cohort:

   Inclusion Criteria:
   * Age ≥18 years;
   * Histologically confirmed invasive breast carcinoma;
   * Clinical stage II-III at presentation;
   * Complete basic information and image data;
   * Have MRI imaging data at baseline and after the first cycle of NAC;
   * Finish the standard NAC treatment and undergo surgery;

   Exclusion Criteria:
   * With chemotherapy contraindications;
   * Multifocal of multicentric lesions;
   * Poor quality of MRI images;
2. For validation cohort:

Inclusion Criteria:

* Age ≥18 years;
* Complete basic information and image data;
* Clinical stage II-III at presentation;
* Scheduled for neoadjuvant chemotherapy;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Signed informed consent;

Exclusion Criteria:

* With chemotherapy contraindications;
* Metastatic breast cancer;
* Multifocal of multicentric lesions;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selection of patients diagnosed with breast cancer and treated with neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity | up to 28 weeks
  Testing the sensitivity of NeoMDSS model to predict pCR using the area under receiver operating characteristic curve.

SECONDARY OUTCOMES:
Specificity | up to 28 weeks
  Testing the sensitivity of NeoMDSS model to predict non-pCR using the area under receiver operating characteristic curve.
Specificity | up to 6 weeks
  Testing the difference in the tumor shrinkage patterns on magnetic resonance imaging (MRI) in triple-negative breast cancer patients receiving neoadjuvant therapy , as well as the correlation between tumor regression pattern and efficacy.

OTHER OUTCOMES:
Shrinkage pattern | up to 28 weeks
  The difference in tumor regression shrinkage patterns between the different treatment groups. Based on the MRI after the first cycle, the tumor SPs were grouped into three categories: CS, diffuse decrease, and no change or enlargement.
correlation between shrinkage patterns and efficacy | up to 28 weeks
  The correlation between tumor regression shrinkage patterns and treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Kun, MD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zou J, Zhang L, Chen Y, Lin Y, Cheng M, Zheng X, Zhuang X, Wang K. Neoadjuvant Chemotherapy and Neoadjuvant Chemotherapy With Immunotherapy Result in Different Tumor Shrinkage Patterns in Triple-Negative Breast Cancer. J Breast Cancer. 2024 Feb;27(1):27-36. doi: 10.4048/jbc.2023.0136. Epub 2023 Nov 17. PMID 37985386